CLINICAL TRIAL: NCT03627481
Title: Sleep Quality After Nasosinusal Surgery in AERD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Marcos Alejandro Jimenez Chobillon, Professor, Instituto Nacional de Enfermedades Respiratorias
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C34-18
Record Dates: First submitted 2018-07-04; First posted 2018-08-13 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Aspirin-exacerbated Respiratory Disease; Sleep
Keywords: endoscopic sinus surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AERD patients (Experimental): Patients managed with Endoscopic sinus surgery for treatment of AERD.
  Interventions: Procedure: Endoscopic sinus surgery

INTERVENTIONS:
Procedure: Endoscopic sinus surgery — Endoscopic sinus surgery for nasal polyposis

SUMMARY:
Aspirin exacerbated respiratory disease presents as a triad composed by asthma, eosinophilic rinosinusitis and intolerance to aspirin and NSAIDS. In subjects with chronic rhinosinusitis sleep alterations have been found, with important improvement after surgery, but those alterations and improvements have not been studied in patients diagnosed with AERD who, due to their comorbidities, may present more severe pre surgical symptoms and a more important post-surgical improvement. The investigators aim to study patients with AERD sleep, quality of life and symptoms before surgery, and one, three and six months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* AERD patients.
* Cumbersome nasal polyposis with poor treatment response

Exclusion Criteria:

* Previously diagnosed sleep disorder.
* Psychiatric disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep quality assessed by the Pittsburgh sleep quality index. | 6 months
  Total score in Pittsburgh sleep quality index, basal and after surgery. Total score in Pittsburgh sleep quality index, before and after surgery. The Pittsburgh sleep quality index has a global score in which a higher score indicates a worse sleep quality, with a global score higher than five differentiating those with good and bad sleep quality. In order to obtain the global score, individual questions are grouped in seven components, to which a 0 to 3 score is assigned and all components scores are added. The total range of the global score goes from 0 to 21.

SECONDARY OUTCOMES:
Objective sleep quality assessed by actigraphy. | Basal; 3 and 6 months
  Sleep efficiency as measured by actigraphy (worn for one week), basal and after. Efficiency is calculated as the average of eficiency for each night.
Quality of life assessed by the Asthma Quality of Life Questionnaire | Basal; 1, 3 and 6 months
  Evaluated with the Asthma Quality of Life Questionnaire, basal and after surgery. The questionnaire has 32 questions with four areas or dominions (activity limitations, asthma symptoms, emotional state and ambient exposition), each question is scored from 1 to 7, with 1 being maximum affectation and 7 no affectation. Final score for each area is obtained by averaging the score for the corresponding questions.
Nasal symptoms assessed by the SNOT - 22 | Basal; 1, 3 and 6 months
  Change in nasal symptoms evaluated via the SNOT 22 questionnaire, basal and after surgery. The sino-nasal outcome test (SNOT-22). This questionnaire is composed by 22 questions that are answered from 0 to 5, with 0 defining no burden and 5 maximal burden, with a total score range from 0 to 110, with a higher score indicating worse symptoms. The total score is obtained by adding the individual question scores.
Asthma symptoms assessed by the Asthma Control Test. | Basal; 1, 3 and 6 months
  Changes on symptoms as evaluated by the score on Asthma Control Test, basal and after surgery. The asthma control test (ACT) has five questions that are answered with scores from 1 to 5, with a total score (obtained by adding the individual question score) from 5 to 25. A higher score indicates worse asthma control. A total score of 19 is considered a cut point for uncontrolled patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided